CLINICAL TRIAL: NCT00898573
Title: Study of Resistance Mechanisms Against Lapatinib in Patients With ErbB-2-Positive Breast Cancers
Brief Title: Lapatinib Resistance in Patients With Breast Cancer
Status: Withdrawn | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE15107; P30CA043703 (NIH); CASE15107 (Other: Case Comprehensive Cancer Center); CASE-15107-CC488
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Cell Separation; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Previously collected tumor tissue samples are obtained for genetic analysis studies. Patients also undergo blood sample collection for extraction of DNA.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lapatinib ditosylate
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: cell sorting
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about cancer and the development of drug resistance in patients.

PURPOSE: This research study is looking at lapatinib resistance in patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify secondary ErbB2 mutations in tumor tissue samples from patients with ErbB2-positive breast cancer treated with lapatinib ditosylate.
* To investigate ErbB2 copy number changes and expression levels.
* To determine abnormalities of other pathways (e.g., c-MET and PI3K) as potential mechanisms of resistance.

OUTLINE: Previously collected tumor tissue samples* are obtained for genetic analysis studies. Samples are analyzed for secondary ErbB2 mutations by nested PCR; ErbB2 copy number changes by quantitative PCR and standard histological FISH; and ErbB2 expression levels by quantitative RT-PCR and IHC. Patients also undergo blood sample collection for extraction of DNA (as normal control DNA) and isolation of EpCAM-positive circulating tumor cells using immunomagnetic cell separation technology. Additional research studies may include mutational and amplification analysis of the c-MET and PI3K pathways.

NOTE: *Patients may undergo biopsy if a post-treatment tumor tissue sample is unavailable.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed invasive breast cancer

  * ErbB2-positive disease
* Has received or is currently receiving lapatinib ditosylate

  * Documented clinical benefit while receiving lapatinib ditosylate (e.g., stable disease of ≥ 12 weeks duration OR a radiographic response)
* Must have tumor tissue samples available for research studies
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Not pregnant*
* Coagulation profile normal*
* Platelet count > 100,000/mm³* NOTE: *For patients requiring a post-treatment biopsy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent chemotherapy or trastuzumab (Herceptin®) allowed
* No concurrent anticoagulants, including warfarin or low-molecular weight heparin*
* No concurrent antiplatelet therapy, including aspirin, clopidogrel, or other antiplatelet agents* NOTE: *For patients requiring a post-treatment biopsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07

PRIMARY OUTCOMES:
Secondary ErbB2 mutations
ErbB2 copy number changes and expression levels
Abnormalities of other pathways (e.g., c-MET and PI3K) as potential mechanisms of resistance

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Budd, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Balazs Halmos, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (9):
- United States (9):
  - Geauga Regional Hospital, Cleveland, Ohio
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Cleveland, Ohio